CLINICAL TRIAL: NCT02761603
Title: Autonomic and Immuno-Vascular Mechanisms of Antihypertensive Effects of Tai Chi
Brief Title: Healthy Aging Practice-centered Instruction Cardiovascular Health Investigation (HAPI-CHI)
Acronym: HAPI-CHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Laura S. Redwine, PhD, Asst Adjunct Prof, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01HL126056 (NIH)
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Hypertension; Prehypertension
MeSH Terms: conditions — Hypertension; Prehypertension | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Aging Practice-centered Instruction (HAPI) (Active Comparator): 24 hours of group instruction in which experts present on a variety of health-related topics followed by class discussion, goal-setting, and goal review. Themes will include: sleep, nutrition, mental health, social support, bone-health, diabetes prevention, cognitive wellness, and resilience.
  Interventions: Behavioral: Healthy Aging Practice-centered Instruction (HAPI)
- Tai Chi (CHI) (Experimental): 24 hours of group instruction in 8 meditative Tai Chi movements.
  Interventions: Behavioral: Tai Chi (CHI)

INTERVENTIONS:
Behavioral: Healthy Aging Practice-centered Instruction (HAPI) — Sessions will include interactive activities derived from the CDC's "Program to Encourage Active and Rewarding LiveS (PEARLS)" and will include lectures based on health-related topics from presentations given by experts as part of the UC San Diego Stein Institute of Aging's Successful Aging project. The PEARLS Problem Solving Treatment (PST) group discussions will be facilitated by a trained instructor in order for participants to identify problems or barriers they have in engaging in healthy behaviors relevant to each of 12 topic areas (e.g. sleep, nutrition, mental health, social support, bone health, diabetes prevention, cognitive wellness, and resilience). Each session will be composed of: Successful Aging video (45 min), discussion (40 min), and identifying problem solving strategies (25 min) with a homework assignment each week, for a total of 24 hours of in-class instruction and discussion.
  Arms: Healthy Aging Practice-centered Instruction (HAPI)
Behavioral: Tai Chi (CHI) — Sessions will include expert instruction in the brief Yang-style 8-form Tai Chi meditative movements. Each class will include a 10-minute warm-up and cool-down plus 40 minutes of Tai Chi instruction and or practice, for a total of 24 hours of in-class instruction
  Arms: Tai Chi (CHI)

SUMMARY:
Over 30% of American adults have hypertension (HTN) (high blood pressure), and the rate increases considerably with age; 64% of men and 78% of women over 65 have HTN. High blood pressure associated with HTN can force of the blood against artery walls with enough pressure that it can eventually cause health problems, such as heart disease and stroke. HTN is one of the most significant causes of early death worldwide and one of the most preventable causes of death. Many studies reveal that lowering blood pressure (BP) reduces the incidence of diseases of the heart and blood vessels. Non-drug related treatments are known to reduce BP which can have a great effect on public health. Research suggests that Tai Chi (TC) is effective in lowering BP in patients with HTN, but because of the low quality of existing studies there is no definite proof. Also, it is not known how TC reduces BP. One possibility is that TC practice, which is shown to reduce psychological distress such as anxiety and depression and reduce the body's responses to stress, can improve the balance of the autonomic nervous system (the part of your nervous system that controls beating of the heart and the widening or narrowing of blood vessels). This may lead to lower BP. The investigators plan to investigate the pathways among autonomic, blood vessel, immune and psychological factors in relation to BP changes in response to 12-weeks of TC compared with Healthy Aging Practice-centered Education (HAP-E). 250 older adults (60+ years old) with mild HTN will be enrolled, and the investigators will take several measurements of heart and nervous system functioning. The investigators hypothesize that performing TC for 12 weeks will result in autonomic "re-regulation" which will improve BP and blood vessel health (Aim 1) and sympathetic nervous system (part of the nervous system that serves to speed up heart rate, contract blood vessels, and raise blood pressure) regulation of the immune system (Aim 2). Lastly, the investigators hypothesize that psychological factors will be related to TC effects on autonomic regulation (Aim 3). Findings from the investigators study will hopefully shed light on the pathways by which TC reduces BP. Also, the particular effects of TC ("meditative movement") in an older, "hard-to-treat" hypertensive population will be better understood.

ELIGIBILITY:
Inclusion Criteria:

1. 1. SBP≥130 but overall BP ≤ 170/110;
2. Able to perform light to moderate exercise;
3. Able to give informed consent;
4. Able to complete study assessments as described;
5. Understand study procedures and to comply with them for the entire length of the study;
6. 5. 60+ years;
7. Able to complete written questionnaires without assistance (reading devices okay);
8. Have not had a fall in that resulted in hospitalization in the past 12 months;
9. Willing to be randomized to TC or HAP-E;
10. Able to attend regular study activities at the center and/or UCSD.

Exclusion Criteria:

1. Currently performing meditation for more than 15 minutes at a time 2X/week or more);
2. Currently performing moderate exercise (enough to work up a sweat) for more than 15 minutes 2X/week or more.
3. Oxygen-dependent COPD;
4. Stroke, cerebral neurologic impairment, cardiac surgery or MI within the past year;
5. Current use of mood stabilizers, or antipsychotics;
6. Medications (steroids) and conditions affecting our immune assays or our physiological measures of vascular function (anti-cholinergics);
7. Severe kidney disease;
8. Current cancer diagnosis or treatment;
9. Insulin-dependent diabetes mellitus;
10. Meets criteria for bipolar disorder, schizophrenia, substance use disorder;
11. Suicidality;
12. Inability to read and write in English;
13. Inability to provide written informed consent;
14. Inability to adequately answer questions on the post-consent assessment;
15. Current smoker;
16. Body Mass Index > 40 kg/m2;
17. Currently meets criteria for major depressive episode (per patient self-report of clinical diagnosis by a professional);

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-04; Primary Completion 2021-05 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in Blood Pressure (mmHg)

SECONDARY OUTCOMES:
Stroke Volume | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in Stroke Volume (mL)
Cardiac Output | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in Cardiac Output (mL/min)
Total Peripheral Resistance (TPR) | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in TPR (mmHg·min/l)
Ejection Fraction (EF) | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in EF (%)
Pulse Wave Velocity (PWV) | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in PWV
Heart Rate Variability (HRV) | Pre- to post-intervention (12 weeks)
  Change From Pre-intervention to Post-intervention in HRV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kohn JN, Lobo JD, Troyer EA, Wilson KL, Ang G, Walker AL, Pruitt C, Pung MA, Redwine LS, Hong S. Tai chi or health education for older adults with hypertension: effects on mental health and psychological resilience to COVID-19. Aging Ment Health. 2023 Mar;27(3):496-504. doi: 10.1080/13607863.2022.2053836. Epub 2022 Mar 21. PMID 35311437